CLINICAL TRIAL: NCT05886855
Title: Evaluation of PerioMonitor for Detection of Oral Inflammatory Load (OIL) in Human Subjects.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Oral Science International Inc. (Industry)
Collaborators: Advarra (Industry)
Responsible Party: Sponsor
Other Study IDs: 230123-01
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Oral Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PerioMonitor Testing: 400 Subject to be tested for Oral Inflammatory Load (OIL) with PerioMonitor. Same subjects to be tested for Oral Inflammation with the BOP method and neutrophil count.

SUMMARY:
The purpose of this multicenter, prospective, single arm Study is to evaluate the efficacy and safety of PerioMonitor as an aid to the detection of oral inflammation associated with periodontal diseases.

PerioMonitor is an IVD device for the rapid, semi-quantitative detection of neutrophil enzyme activity in oral samples. This test is intended for prescription use at Point-of-Care ("POC") settings by health care professionals.

DETAILED DESCRIPTION:
The purpose of this multicenter, prospective, single arm Study is to evaluate the efficacy and safety of PerioMonitor as an aid to the detection of oral inflammation associated with periodontal diseases.

PerioMonitor is an IVD device for the rapid, semi-quantitative detection of neutrophil enzyme activity in oral samples. This test is intended for prescription use at Point-of-Care ("POC") settings by health care professionals.

The primary objective of this Study is to evaluate the Positive Percent Agreement (PPA)PPA and the Negative Percent Agreement (NPA)NPA of PerioMonitor for semi-quantitative detection of neutrophil enzyme activity in human oral specimens, to detect oral inflammation associated with periodontal diseases (subjects having more than 50 000 neutrophils/mL in their oral specimen or having more than 10% of bleeding sites when tested with the BOP method).

The secondary objective is to validate the claim that PerioMonitor can be used in POC settings (i.e., representative of the intended users and under conditions similar to the conditions of use), at the time of the consultation, with instant availability of results, by healthcare professionals (HCP) working in a dental clinic (i.e. with the background, education, and training of those who will perform the test in its intended environment) that are not qualified laboratory technicians, to make immediate and informed decisions about patient care.

ELIGIBILITY:
Inclusion Criteria:

* subject > 18 years old;
* subject fluent in English; and
* subject has signed the ICF

Exclusion Criteria:

* Subject with altered mental status/inability to provide informed consent or follow the procedure of the Study; and
* Subject using immunosuppressants including biologics such as adalimumab (Humira) and infliximab (Remicade); or calcineurin inhibitors such as tacrolimus (Envarsus XR or Protopic) and cyclosporine (Gengraf, Neotal or Sandimmmune); or corticosteroids (Prednisone); or azathioprine (Imuran)
* Oral rinse specimens received 5 days or more after PerioMonitor testing by the clinical laboratory
* Previous enrolment into the current Study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals visiting a dental clinic for a regular exam.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-05-24 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Bleeding on Probing (BOP) | 6 months
  Confirmation of oral inflammation if BOP is equal or above 10%

IPD SHARING:
Plan to Share IPD: No